CLINICAL TRIAL: NCT01625988
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients With Migraine
Brief Title: A Study of LY2951742 in Participants With Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART-01; ART-01 (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2014-04

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2951742 (Experimental): LY2951742: 150 milligrams (mg), subcutaneous (SC) injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
  Interventions: Drug: LY2951742
- Placebo (Placebo Comparator): Placebo: 0.9% Sodium Chloride, Untied States Pharmacopoeia (USP), subcutaneous (SC) injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2951742
  Arms: LY2951742
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of LY2951742 in the prevention of migraine headache in migraineurs with or without aura during 3 months of treatment.

DETAILED DESCRIPTION:
The study is comprised of 4 trial periods:

1. Screening and washout (5-45 days)
2. Baseline for assessment of the type, frequency, and severity of headaches (28-38 days)
3. Treatment (12 weeks)
4. Follow-up (12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Have a history of migraine as defined by the International Headache Society (IHS) International Classification of Headache Disorders II guidelines 1.1 and 1.2 (ICHD-II, Cephalgia 2004) of at least 1 year prior to enrollment, migraine onset prior to age 50, and a moderate frequency of migraine headaches
* Women of child-bearing potential (not surgically sterile or at least 1 year post-menopause) must test negative for pregnancy at the time of screening based on a serum pregnancy test and must agree to use a reliable method of birth control during the study and for 3 months following completion of participation in the study
* Have clinical laboratory test results within normal reference ranges or, if outside the normal range, judged not clinically significant by the Investigator
* Must not be on any migraine prevention therapy, including botulinum toxin (Botox)
* Agree not to post any personal medical data related to the study or information related to the study on any website or social media site (for example, Facebook, Twitter, et cetera) until the trial has completed

Exclusion Criteria:

* Current enrollment in, or discontinuation within the last 30 days from, a clinical trial involving any investigational drug or device, or concurrent enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study
* Previous completion or withdrawal from this study or any other study investigating LY2951742 or other therapeutic antibodies that target calcitonin gene-related peptide (CGRP)
* History of chronic migraine or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and basilar-type migraine
* History of headache (for example, cluster headache or Medication Overuse Headache [MOH]) other than migraine or tension type headache as defined by IHS ICHD-II within 12 months prior to randomization
* Evidence of significant active psychiatric disease including, but not limited to, manic depressive illness, schizophrenia, generalized anxiety disorder, obsessive compulsive disorder, personality disorders, or other serious mood, anxiety, depression, or substance use disorders
* Have a history or presence of any other medical illness that in the judgment of the Investigator, indicates a medical problem that would preclude study participation
* Women who are pregnant or nursing
* Confirmed corrected QT (QTc) interval >470 milliseconds (msec) for women and >450 for men
* Excessive alcohol, opiate, or barbiturate use; history of drug abuse or dependence
* In the opinion of the Investigator, have no other issues that would interfere with compliance with the study requirements and completion of evaluations required for this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2012-06-28 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (37):
  - Neurological Physicians of Arizona / Clinical Research Advantage, Gilbert, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Mayo Foundation for Medical Education and Research - Mayo Clinic, Scottsdale, Arizona
  - PRI Encino, Encino, California
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - Collaborative Neuroscience Network Inc., Long Beach, California
  - PRI Los Alamitos, Los Alamitos, California
  - PRI Newport Beach, Newport Beach, California
  - Medical Center for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - University of California, San Francisco (UCSF) Medical Center - Headache Center, San Francisco, California
  - California Medical Clinic for Headache Inc, Santa Monica, California
  - Radiant Research - Denver, Denver, Colorado
  - Florida Clinical Research Center LLC, Maitland, Florida
  - Accelovance, Inc, Melbourne, Florida
  - Renstar Medical Research, Ocala, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Neurology Clinical Research Inc, Sunrise, Florida
  - MedVadis Research, Watertown, Massachusetts
  - Westside Family Medical Center, PC, Kalamazoo, Michigan
  - Ryan Headache Center, St. John's Mercy Medical Group, Chesterfield, Missouri
  - Clinvest, A Division of Banyan Group, Inc., Springfield, Missouri
  - Prarie Fields Medicine/Clinical Research Advantage, Fremont, Nebraska
  - James Meli DO Ltd (Clinical Research Advantage), Henderson, Nevada
  - Clinical Research Advantage, Henderson, Nevada
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - PMG Research of Bristol, Bristol, Tennessee
  - ClinSearch, Chattanooga, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee
  - FutureSearch Trials of Neurology and Sleep Lab, Austin, Texas
  - Neurology Studies of Austin, A Division of DermResearch Inc., Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Clinical Trial Network (CTN Texas), Houston, Texas
  - Neurology & Headache Treatment Center, McLean, Virginia

REFERENCES:
- [Derived] Stauffer VL, Turner I, Kemmer P, Kielbasa W, Day K, Port M, Quinlan T, Camporeale A. Effect of age on pharmacokinetics, efficacy, and safety of galcanezumab treatment in adult patients with migraine: results from six phase 2 and phase 3 randomized clinical trials. J Headache Pain. 2020 Jun 23;21(1):79. doi: 10.1186/s10194-020-01148-9. PMID 32576229
- [Derived] Goadsby PJ, Dodick DW, Martinez JM, Ferguson MB, Oakes TM, Zhang Q, Skljarevski V, Aurora SK. Onset of efficacy and duration of response of galcanezumab for the prevention of episodic migraine: a post-hoc analysis. J Neurol Neurosurg Psychiatry. 2019 Aug;90(8):939-944. doi: 10.1136/jnnp-2018-320242. Epub 2019 Apr 19. PMID 31004075
- [Derived] Dodick DW, Goadsby PJ, Spierings EL, Scherer JC, Sweeney SP, Grayzel DS. Safety and efficacy of LY2951742, a monoclonal antibody to calcitonin gene-related peptide, for the prevention of migraine: a phase 2, randomised, double-blind, placebo-controlled study. Lancet Neurol. 2014 Sep;13(9):885-92. doi: 10.1016/S1474-4422(14)70128-0. Epub 2014 Aug 10. PMID 25127173

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: 0.9% Sodium Chloride, Untied States Pharmacopoeia (USP), SC injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
Period: Overall Study
Arm/Group | LY2951742 | Placebo
Started | 108 (One participant was randomized inappropriately and was discontinued before start of study treatment.) | 110
Received at Least One Dose of Study Drug | 107 | 110
Completed | 94 | 97
Not Completed | 14 | 13
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Randomized Inappropriately | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo: 0.9% Sodium Chloride, USP, SC injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
- Total: Total of all reporting groups
Arm/Group | LY2951742 | Placebo | Total
Number analyzed (Participants) | 107 | 110 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All participants who received at least one dose of study drug and had baseline Age data.
  years
    number analyzed (Participants) | 107 | 109 | 216
    (all) | 40.9 (11.4) | 41.9 (11.7) | 41.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 96 | 184
  Male | 19 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 96 | 97 | 193
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 25 | 26 | 51
  White | 76 | 74 | 150
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 107 | 110 | 217

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Number of Migraine Headache Days in the Last 28-day Period of the 12-week Treatment Phase
Description: The criteria for a migraine headache was adapted from the standard International Headache Society (IHS) International Classification of Headache Disorders II guidelines 1.1 and 1.2 (ICHD-II, Cephalgia 2004). The definition of a migraine headache was a headache with or without aura, of ≥30 minutes (min) duration, and with both ("A" and "B") required features from the IHS ICHD-II definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia. Least square (LS) means were calculated using mixed model repeated measures (MMRM) with baseline value, treatment, month, and treatment-by-month interaction as fixed effects and participant as random effect.
Time Frame: Baseline, 12 weeks
Population: All participants with a valid 28-day baseline assessment of migraine headache days who received at least 1 dose of study treatment and had evaluable postbaseline headache data.
Measure: Least Squares Mean (Standard Error); unit: Migraine headache days
Arm/Group | LY2951742 | Placebo
Number analyzed (Participants) | 106 | 110
Migraine headache days | -4.2 (0.30) | -3.0 (0.29)

2. Secondary Outcome: Mean Change From Baseline in the Number of Headache Days in the Last 28-day Period of the 12-week Treatment Phase
Description: Number of calendar days on which a headache lasts ≥4 hours which includes migraines, probable migraines (PM) and nonmigraines. Criteria for migraine headache (MH) was adapted from standard IHS ICHD-II guidelines 1.1 and 1.2 (Cephalgia 2004). Definition of MH was headache with or without aura, of ≥30 min duration, and with both ("A" and "B") required features from IHS ICHD-II definition. Required feature "A" includes ≥2 of following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of following during headache: nausea and/or vomiting, or photophobia and phonophobia. PM is headache with or without aura, but missing 1 feature needed to fulfill all criteria for MH. LS means were calculated using MMRM with baseline value, gender, treatment, month, and treatment-by-month interaction as fixed effects and participant as random effect.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Headache days
Arm/Group | LY2951742 | Placebo
Number analyzed (Participants) | 106 | 110
Headache days | -4.9 (0.40) | -3.7 (0.40)

3. Secondary Outcome: Mean Change From Baseline in the Number of Migraine Attacks in the Last 28-day Period of the 12-week Treatment Phase
Description: A migraine attack was defined as beginning on any day a migraine headache day was recorded and ending when a migraine headache-free day occurred. The criteria for a migraine headache was adapted from the standard IHS ICHD-II guidelines 1.1 and 1.2 (Cephalgia 2004). The definition of a migraine headache was a headache with or without aura, of ≥30 minutes duration, and with both ("A" and "B") required features from the IHS ICHD-II definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia. LS means were calculated using MMRM with baseline value, gender, treatment, month, and treatment-by-month interaction as fixed effects and participant as random effect.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Migraine attacks
Arm/Group | LY2951742 | Placebo
Number analyzed (Participants) | 106 | 110
Migraine attacks | -3.1 (0.23) | -2.3 (0.24)

4. Secondary Outcome: Percentage of Responders
Description: Percentage of participants with greater than 50% reduction in the number of migraine headache days in a 28-day period. The criteria for a migraine headache was adapted from the standard International Headache Society (IHS) International Classification of Headache Disorders II guidelines 1.1 and 1.2 (ICHD-II, Cephalgia 2004). The definition of a migraine headache was a headache with or without aura, of ≥30 minutes duration, and with both ("A" and "B") required features from the IHS ICHD-II definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia.
Time Frame: Baseline, 4, 8, and 12 weeks
Population: All participants with a valid 28-day baseline assessment of migraine headache days who received at least 1 dose of study treatment and had evaluable postbaseline headache data during the time period of analysis.
Measure: Number; unit: Percentage of participants
Groups:
- LY2951742: LY2951742 (LY): 150 milligrams (mg), subcutaneous (SC) injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
Arm/Group | LY2951742 | Placebo
Number analyzed (Participants) | 107 | 110
Percentage of participants
  Week 4: number analyzed (Participants) | 62 | 41
  Week 4 | 57.9 | 37.3
  Week 8: number analyzed (Participants) | 66 | 47
  Week 8 | 61.7 | 42.7
  Week 12: number analyzed (Participants) | 69 | 47
  Week 12 | 64.5 | 42.7

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- LY2951742 Treatment Period: LY2951742: 150 mg, SC injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
- Placebo Treatment Period: Placebo: 0.9% Sodium Chloride, USP, SC injection on Day 1 and then once every other week for a total of 6 doses during the 12-week Treatment Period.
- LY2951742 Posttreatment Period: LY2951742: The LY2951742 posttreatment period reporting group includes participants who received 150 mg LY2951742, completed the 12-week treatment period, and entered the posttreatment period. The posttreatment period began after Week 12 and lasted up to 12 weeks. Note: participants who discontinued early in the treatment phase did not enter the 12-week posttreatment follow-up period.
- Placebo Posttreatment Period: Placebo: The Placebo posttreatment period reporting group includes participants who received 0.9% Sodium Chloride, USP; completed the 12-week treatment period; and entered the posttreatment period. The posttreatment period began after Week 12 and lasted up to 12 weeks. Note: participants who discontinued early in the treatment phase did not enter the 12-week posttreatment follow-up period.
Arm/Group | LY2951742 Treatment Period | Placebo Treatment Period | LY2951742 Posttreatment Period | Placebo Posttreatment Period
Serious Adverse Events (participants affected / at risk) | 0/107 | 1/110 | 2/98 | 3/103
Other Adverse Events (participants affected / at risk) | 36/107 | 30/110 | 6/98 | 2/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2951742 Treatment Period (N=107) | Placebo Treatment Period (N=110) | LY2951742 Posttreatment Period (N=98) | Placebo Posttreatment Period (N=103)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/88 (0) | 0/96 (0) | 1/80 (1) | 0/90 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/88 (0) | 0/96 (0) | 0/80 (0) | 1/90 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2951742 Treatment Period (N=107) | Placebo Treatment Period (N=110) | LY2951742 Posttreatment Period (N=98) | Placebo Posttreatment Period (N=103)
Nausea (Gastrointestinal disorders) | 4 (4) | 9 (10) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 18 (65) | 7 (14) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 10 (11) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Arteaus Therapeutics executed the contracts and trial, and the Principal Investigators are restricted by any original contractual disclosure restrictions or agreements with Arteaus Therapeutics.